CLINICAL TRIAL: NCT06537089
Title: Comparative Study Between Using WHO Labour Care Guide & Modified WHO Partograph in Reducing Primary Cesarean Section in Primiparous Women in Active First Stage of Labour.
Brief Title: Comparative Study Between Using WHO Labour Care Guide & Modified WHO Partograph
Status: Recruiting | Type: Observational
Sponsor: Hend Mahmoud Abdelghany (Other)
Responsible Party: Sponsor-Investigator, Hend Mahmoud Abdelghany, Lecturer of Obstetrics and Gynecology, Cairo University, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Other Study IDs: MD-400-2023
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Labor Onset and Length Abnormalities; 37 or More Completed Weeks of Gestation; First Birth
Keywords: labour Monitoring; primiparous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This randomized clinical trial is based on comparing the efficiency of modified WHO partographs vs. the new WHO labour care guide in monitoring and assessing the outcome of labour.

DETAILED DESCRIPTION:
A group of primiparous women in first stage of labour will be randomized into two groups then monitored during first stage of labour. First group will be monitored by modified WHO partograph. The rest of participants will be monitored by WHO labour care Guide. The labour will be monitored regarding progress rate, mode of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Primiparous women.
* Term gestation between 37 and 40 weeks.
* Maternal age from 18 -35 years
* Body mass index BMI of 18.5 to 29.9 kg/m2
* Cephalic presentation. 6. Active first stage of labour

Exclusion Criteria:

* Women with any medical comorbidities, such as (hypertension, diabetes mellitus, renal disease, or pulmonary disease).
* Women with presence of any obstetrical complications, such as preterm birth, multiple gestation, breech presentation, postdated pregnancy, or bad obstetrical history.
* women who were given intrapartum epidural analgesia.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This randomized controlled study will be conducted on 230 low-risk pregnant women admitted in labor in the labor room (LR) in kasr Alainy hospital.
  Enrollment at the time of admission as per inclusion and exclusion criteria. After informed consent, randomization and allocation to study and control groups will be conducted using a computer- generated sequence, and enrollment continues until the desired sample size of 115 is reached in each group.
Sampling Method: Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of primary caesarean section | First and second stage of labour
  number of women will undergo Caesarean section after monitoring, whether by Modified WHO partograph or a labour care Guide

SECONDARY OUTCOMES:
Duration of active phase of first stage of labour | First stage of labour
Duration of second stage of labour | Second stage of labour
need for oxytocin use | First stage of labour

CONTACTS AND LOCATIONS:
Locations (1):
- kasr Al Aini, Faculty of Medicine, Cairo University, Cairo, Old Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided